CLINICAL TRIAL: NCT05400668
Title: The Reliability and Validity of the Turkish Version of the Medial Tibial Stress Syndrome (MTSS-Tr) Score
Brief Title: The Turkish Version of the Medial Tibial Stress Syndrome Score
Status: Completed | Type: Observational
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Merve Demir Benli, Medical Doctor, Sports Medicine Physician, Bozyaka Training and Research Hospital
Other Study IDs: mdbenli
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Medial Tibial Stress Syndrome
MeSH Terms: conditions — Medial Tibial Stress Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The medial tibial stress syndrome (MTSS) score was originally developed in Dutch to assess severity of disease relative to patient-reported outcome, particularly patients with MTSS. The purpose of this study was to translate and cross-culturally adapt the MTSS score into Turkish and investigate its psychometric properties.

DETAILED DESCRIPTION:
The medial tibial stress syndrome (MTSS) score was originally developed in Dutch to assess severity of disease relative to patient-reported outcome, particularly people with MTSS. The purpose of this study was to translate and cross-culturally adapt the MTSS score into Turkish and investigate its psychometric properties. Fourty-eight individuals with MTSS will include. Within a 7-day period after the first assessment, the participants completed the Turkish version of the MTSS score to evaluate test-retest reliability.

Cronbach's alpha (α) was used to assess internal consistency. Construct validity was examined total score of PCS domain of SF-36-Tr with MTSS-Tr total score in the first visit. Concurrent validity was examined by evaluating the relationship between pain level and Detmer's classification with MTSS score in the first visit. The pain level of the patient assessed with visual analog scale (VAS) score.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with MTSS by a sports medicine physician
* Patients aged between 18 and 75 years
* Patients whose native language is Turkish
* Patients who volunteered to participate in the study

Exclusion Criteria:

* Having tibia fracture history,
* Patients with suspected stress fracture or chronic compartment syndrome,
* Pregnant and breastfeeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include 48 patients diagnosed with medial tibial stress syndrome (MTSS) by the sports medicine physicians in İzmir Bozyaka Training and Research Hospital, Tepecik Training and Research Hospital and Ege University. The individuals who volunteers and meets the inclusion criteria will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-10-13 (Actual)

PRIMARY OUTCOMES:
Medial Tibial Stress Syndrome Score | Baseline (First assessment)
  The MTSS total score is a reliable and valid tool to assess severity in patient with MTSS. The 14-item MTSS score was designed to assessing limitations in sporting activities, pain while performing sporting activities, pain while performing activities of daily living and pain at rest. Items have four response options with descriptors for each response category. Higher item scores indicate a more severe pain or limitation and hence more severe MTSS symptoms. Participants were asked to fill out the MTSS score with their most painful shin in mind, in case of bilateral symptoms.

SECONDARY OUTCOMES:
Medial Tibial Stress Syndrome Score | Within a 7-day period after the first assessment (Second assessment)
  The MTSS total score is a reliable and valid tool to assess severity in patient with MTSS. The 14-item MTSS score was designed to assessing limitations in sporting activities, pain while performing sporting activities, pain while performing activities of daily living and pain at rest. Items have four response options with descriptors for each response category. Higher item scores indicate a more severe pain or limitation and hence more severe MTSS symptoms. Participants were asked to fill out the MTSS score with their most painful shin in mind, in case of bilateral symptoms.
36-Item Short Form Survey (SF-36) | Baseline (First assessment)
  The SF-36 is widely used to measure a variety of domains, including pain and limitations while performing activities of daily living, and also in musculoskeletal and sports medicine-related research. Short Form Health Survey (SF-36), which includes two main domains, the physical component score (PCS) and the mental component score (MCS), has been widely used worldwide in studies to assess the health status burden of people and consists of 36 questions that are clustered to yield eight health status scales: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, mental health, reported health transition. The total score of PCS and MCS from 0 to 100, with higher scores indicating higher levels of function and/or better health.
MTSS clinical classification (Detmer's classification) | Baseline (First assessment)
  Physical examination evaluates the localization of pain at the posteromedial edge of tibia. According to the MTSS classification created by Detmer et al.; it is classified as Type 1 in the presence of tenderness only on the tibia, Type 2 in the posteromedial of the tibia at the junction of the periosteum and fascia, and Type 3 in the presence of tenderness in the deep compartment muscles of the posterior tibia.
Evaluating the applicability of the questions | Within a 7-day period after the first assessment (Second assessment)
  Participants evaluate the MTSS questionnaire with additional three Likert-type questions in the first assessment. In the continuation of these questions, there is also a comment section about the simplicity of filling out the survey and the convenience and usefulness of this survey.
Visual Analog Scala (VAS) | Baseline (First assessment)
  Pain is graded from 0 to 10 by Visual Analog Scala (VAS). 0 indicates the least pain and 10 the most pain. The patient gives a value on this scale for the pain she/he feels.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Demir Benli, MD, Study Director — Bozyaka Training and Research Hospital
Locations (1):
- Tepecik Training and Research Hospital, Izmir, Turkey (Türkiye)

REFERENCES:
- [Derived] Demir Benli M, Winters M, Arslan AS, Ceylan E, Benli C, Ergun M. Validity and Reliability of the Turkish Version of the Medial Tibial Stress Syndrome Score. Orthop J Sports Med. 2024 Dec 5;12(12):23259671241296885. doi: 10.1177/23259671241296885. eCollection 2024 Dec. PMID 39640185